CLINICAL TRIAL: NCT05510869
Title: Comparison of Surgically Induced Astigmatism After Microincision Cataract Surgery (B-MICS 1.4 mm and C-MICS 1.8 mm) and C- SICS 2.4 mm
Brief Title: Evaluation of the Impact of Corneal Width on Surgically Induced Astigmatism (SIA) and Functional Results After Bimanual 1.4 mm Microincision Cataract Surgery (B-MICS), Coaxial 1.8 mm MICS (C-MICS) and 2.4 mm Small Incision Cataract Surgery (C-SICS).
Acronym: MICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Magdalena Kucharczyk-Pośpiech, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNN/230/13/KE
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Cataract; Corneal Astigmatism; Corneal Incision Contracture
Keywords: surgically induced astigmatism; phacoemulsification; bimanual microincision cataract surgery; coaxial microincision cataract surgery; small incision cataract surgery; clear corneal incision
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B-MICS 1.4 mm (Experimental): bimanual 1.4 mm cataract surgery (B-MICS)
  Interventions: Procedure: Bimanual 1.4 mm microincision cataract surgery (B-MICS) with IOL implantation in a "wound-assisted" technique. In bimanual MICS group a self-sealing 1.4 mm wide incision was created supratemporally
- C-MICS 1.8 mm (Active Comparator): coaxial 1.8 mm cataract surgery (C-MICS)
  Interventions: Procedure: Coaxial 1.8 mm microincision cataract surgery (C-MICS) with IOL implantation with an injector through the 1.8 mm wide incision created temporally.
- C-SICS 2.4 mm (Active Comparator): coaxial 2.4 mm small incision cataract surgery (C-SICS)
  Interventions: Procedure: Coaxial 2.4 mm small incision cataract surgery (C-SICS) with IOL implantation with an injector through the 2.4 mm wide incision located temporally.

INTERVENTIONS:
Procedure: Bimanual 1.4 mm microincision cataract surgery (B-MICS) with IOL implantation in a "wound-assisted" technique. In bimanual MICS group a self-sealing 1.4 mm wide incision was created supratemporally — microincision cataract surgery (phacoemulsification) with implantation of a foldable, acrylic, hydrophilic IOL Incise® MJ14, Bausch & Lomb
  Arms: B-MICS 1.4 mm
Procedure: Coaxial 1.8 mm microincision cataract surgery (C-MICS) with IOL implantation with an injector through the 1.8 mm wide incision created temporally. — microincision cataract surgery (phacoemulsification) with implantation of a foldable, acrylic, hydrophilic IOL Incise® MJ14, Bausch & Lomb
  Arms: C-MICS 1.8 mm
Procedure: Coaxial 2.4 mm small incision cataract surgery (C-SICS) with IOL implantation with an injector through the 2.4 mm wide incision located temporally. — small incision cataract surgery (phacoemulsification) with implantation of a foldable, acrylic, hydrophilic IOL Incise® MJ14, Bausch & Lomb
  Arms: C-SICS 2.4 mm

SUMMARY:
The aim of the study is to compare functional results and complications of 3 methods of cataract phacoemulsification: bimanual 1.4 mm cataract surgery (B-MICS), coaxial 1.8 mm cataract surgery (C-MICS) and coaxial 2.4 mm small incision cataract surgery.

DETAILED DESCRIPTION:
Reduction of the width of the corneal incision was one the main changes taking place in cataract surgery in recent years. The common use of foldable intraocular lenses (IOLs) and technological development of phaco machines allowed to reduce clear corneal incision below 3 mm. Term of Microincision Cataract Surgery (MICS) understood as cataract phacoemulsification performed with the incision width below 2 mm was defined by professor Alio in 2003. However, despite various modifications introduced in recent years, phacoemulsification still causes damage of the tissues that results in surgically induced astigmatism.

Two MICS techniques have been developed: bimanual microincision cataract surgery (B-MICS) and coaxial microincision cataract surgery (C-MICS).

In the bimanual technique cataract phacoemulsification can be performed through the main incision 1.4 mm wide due to the usage of sleeveless phaco tip (without irrigation) and irrigation chopper. The advantage of separation the irrigation from aspiration is improvement of liquid dynamics in the anterior chamber. Moreover, due to the usage of the irrigation chopper, in B-MICS it is possible to lower the mean ultrasound energy.

In coaxial technique MICS phacoemulsification is performed through the incision 1.8 mm wide with usage of phaco tip with a silicon irrigation sleeve.

The aim of the study is to compare functional results and complications of 3 methods of cataract phacoemulsification: bimanual 1.4 mm cataract surgery (B-MICS), coaxial 1.8 mm cataract surgery (C-MICS) and coaxial 2.4 mm small incision cataract surgery. Moreover, this study aimed to evaluate the impact of corneal width on best corrected visual acuity (uncorrected and corrected), surgically induced astigmatism, endothelial cell loss, intraocular pressure, anterior segment of the eye and central retinal thickness.

ELIGIBILITY:
Inclusion Criteria:

* lens opacities which were an indication for cataract surgery and absence of exclusion criteria,
* cataract sclerosis grade from II to IV in Lens Opacities Classification System LOCS III scale (The Lens Opacities Classification System III).

Exclusion Criteria:

* history of ocular surgery, ocular trauma,
* congenital ocular malformations, amblyopia,
* corneal disorders (including corneal opacities and scars),
* best corrected visual acuity (BCVA) ≥ 0.9,
* preoperative endothelial cell density <1500 cells/mm2,
* history of uveitis, diabetic retinopathy,
* retinal and macular disorders,
* eventful phacoemulsification
* presence of other diseases that could affect the postoperative visual outcomes.

Ages: 35 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
the best corrected visual acuity | 36 months
  examined with digital Snellen chart, measured in decimal scale
the best uncorrected visual acuity | 36 months
  examined with digital Snellen chart, measured in decimal scale
autorefractometry | 36 months
  measured in diopters (D)
keratometry | 36 months
  measured in diopters (D)
intraocular pressure (IOP) | 36 months
  measured in millimeters of mercury (mmHg)
endothelial cell density (ECD) | 36 months
  measured in endothelial cells/mm2
central corneal thickness (CCT) | 36 months
  measured with Anterior Segment Optical Coherence Tomography (AS-OCT), unit of measure: µm (micrometers).
peripheral temporal corneal thickness | 36 months
  measured at the main incision site with Anterior Segment Optical Coherence Tomography (AS-OCT), unit of measure: µm (micrometers)
peripheral nasal corneal thickness | 36 months
  measured with Anterior Segment Optical Coherence Tomography (AS-OCT), unit of measure: µm (micrometers)
anterior chamber depth (ACD) | 36 months
  measured with Anterior Segment Optical Coherence Tomography (AS-OCT) in mm (milimeters).
the white-to-white (WTW) distance - the horizontal corneal diameter | 36 months
  measured with Anterior Segment Optical Coherence Tomography (AS-OCT, unit of measure: mm (milimeters).
length of the clear corneal incision | 36 months
  the chord length measured with Anterior Segment Optical Coherence Tomography (AS-OCT), unit of measure: µm (micrometers)
anterior chamber angle | 36 months
  measured with Anterior Segment Optical Coherence Tomography (AS-OCT) in horizontal scan, unit of measure: degrees
central foveal thickness (CFT) | 36 months
  measured with Optical Coherence Tomography (OCT), unit of measure: µm (micrometers)
parafoveal retinal thickness | 36 months
  measured with Optical Coherence Tomography (OCT), unit of measure: µm (micrometers)

SECONDARY OUTCOMES:
surgically induced astigmatism SIA | 36 months
  measured in dioptres (D) - three different methods were used for calculation of surgically induced astigmatism (SIA): vector analysis method, vector decomposition method (C90), Naeser's polar values method (dKP-90)